CLINICAL TRIAL: NCT00133198
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Clinical Trial Comparing Fixed Doses of 0.25 mg, 0.50 mg and 0.75 mg Pramipexole (Mirapex®) Administered Orally to Investigate the Safety and Efficacy in Patients With Idiopathic Restless Legs Syndrome for 12 Weeks
Brief Title: Efficacy and Safety of Pramipexole Compared to Placebo in the Treatment of Restless Legs Syndrome (RLS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 248.543
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

INTERVENTIONS:
Drug: Pramipexole

SUMMARY:
A 12 week clinical trial was conducted in the United States in order to compare pramipexole (Mirapex®) versus placebo for the ability to reduce the symptoms of restless legs syndrome in adult subjects.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2004-04; Primary Completion 2005-02 (Actual); Study Completion 2005-02

PRIMARY OUTCOMES:
Change from baseline in the total score of RLSRS (Restless Legs Syndrome rating scale for severity) of the IRLSSG (International Restless Legs Syndrome Study Group) | week 12
CGI-I (CGI-Improvement) | week 12

SECONDARY OUTCOMES:
RLSRS response (≥50% reduction from baseline in RLSRS) | at week 4, 6 and 12
CGI-I responder analysis | at week 4, 6 and 12
Change from baseline in CGI-Severity | at week 4, 6 and 12
CGI-therapeutic effect | at week 4, 6 and 12
CGI-Side effects | at week 4, 6 and 12
Patient Global Impression (PGI) | at week 1-4, 6 and 12
Visual analogue scales to assess RLS severity before sleep onset, during night and during day, and satisfaction with sleep | at week 4, 6 and 12
Change from baseline in Epworth sleepiness scale (ESS) | at week 4, 6 and 12
Change from baseline in RLS-QOL (Johns Hopkins Restless Legs Syndrome Quality of Life questionnaire) | at week 6 and 12
Change from baseline in Augmentation Severity Rating Scale of IRLSSG | at week 6 and 12
Change in systolic and diastolic blood pressure (after 5 minutes supine and subsequently after 1 minute standing) | week 12
Change in pulse rate (palpation after 5 minute supine and subsequent after 1 minute standing) | week 12
Change in routine laboratory tests | week 12
Change in Physical examinations including eye examinations with ophthalmoscopic retinal eye examinations and a full skin dermatologic examination | week 12
Change in Electrocardiogram | 12 weeks
Incidence of Adverse evens (including withdrawal symptoms and rebound symptoms) | up to 93 days
Concomitant medication reporting | 12 weeks
Early withdrawal phenomena | 12 weeks
Assessment of sudden onset of sleep (SOOS) | up to 93 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharmaceuticals,Inc./Ridgefield
Locations (44):
- United States (44):
  - Pivotal Research Centers, Peoria, Arizona
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - HealthQuest Clinical Trials Research, San Diego, California
  - Stanford Sleep Clinic, Stanford, California
  - Adult CF Center, Denver, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado
  - CNI Movement Disorders Center, Englewood, Colorado
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - PAB Clinical Research, Brandon, Florida
  - Broward Research Group, Pembroke Pines, Florida
  - Clinical Research Group of St Petersburg, St. Petersburg, Florida
  - Cleveland Clinic Florida- Department of Neurology, Weston, Florida
  - 5671 Peachtree Dunwoody Road, Atlanta, Georgia
  - Atlanta Pulmonary Group, LLC, Atlanta, Georgia
  - Movement Disorders Clinic, Augusta, Georgia
  - Sleepmed, Inc, Macon, Georgia
  - University of Iowa Health Care, Iowa City, Iowa
  - Mid America NeuroScience Institute, Lenexa, Kansas
  - Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - 170 Thomas Johnson Dr, Suite 100, Frederick, Maryland
  - Sleep Health Centers, Newton Center, Massachusetts
  - Henry Ford Hospital - Sleep Disorders and Research Center, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Sleep Disorders Center, Jackson, Mississippi
  - Sleep Medicine Center, St Louis, Missouri
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Winthrop Sleep Disorders Center, Mineola, New York
  - 932 Morreene Road #264, Durham, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wilmington Health Associates, Wilmington, North Carolina
  - Attn: Dr. David Mayleben, Cincinnati, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Attn: Controller/Grants & Contracts Accounting, Oklahoma City, Oklahoma
  - Center For Sleep Medicine, Lafayette Hill, Pennsylvania
  - The Arthritis Group, Philadelphia, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Sleep Associates, Plano, Texas
  - 1500 N. Bearegard St, #300, Alexandria, Virginia
  - Lynchburg Pulmonary Associates, Inc., Lynchburg, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia